CLINICAL TRIAL: NCT01049217
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter Trial Of Pregabalin Versus Placebo In The Treatment Of Neuropathic Pain Associated With HIV Neuropathy (Pregabalin A0081244)
Brief Title: Pregabalin Versus Placebo In The Treatment Of Neuropathic Pain Associated With HIV Neuropathy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A0081244
Record Dates: First submitted 2010-01-13; First posted 2010-01-14 (Estimated); Results first posted 2013-07-17 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2013-08

CONDITIONS: Neuropathy
Keywords: neuropathy; pain; HIV-1; HIV Infections
MeSH Terms: conditions — Pain; HIV Infections | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active drug (Experimental)
  Interventions: Drug: pregabalin
- Control (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: pregabalin — Pregabalin 75 mg-300mg twice daily during the course of the study.
  Arms: Active drug
Drug: placebo — Subjects may be assigned to placebo during this study. The study duration is approximately 19 weeks.
  Arms: Control

SUMMARY:
The purpose of this study is to evaluate the efficacy of pregabalin compared to placebo in reducing neuropathic pain associated with HIV neuropathy.

DETAILED DESCRIPTION:
Based on DMC interim efficacy analysis results indicating a low probability for success the study was terminated on April 2, 2012; the termination was unrelated to any safety findings that could impact patient health.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, ages of 18 or greater
* Documented evidence of HIV-1 infection
* Documented diagnosis of HIV-associated Distal Symmetrical Polyneuropathy (DSP) with subjective sensory symptom of pain
* Pain starts in the feet

Exclusion Criteria:

* Subject has untreated vitamin B12 deficiency (serum B12 level <200 pg/ml) or if treated B12 deficiency -treatment is less than 6 months of B12 supplementation (injection or intranasal B12) prior to screening
* Diabetes mellitus requiring regular medical treatment (other than diet and exercise) or HbA1C >6.9
* Subjects with peripheral neuropathic pain that is not associated with HIV infection; including subjects with conditions such as: Post Herpetic Neuralgia (PHN), Diabetic Peripheral Neuropathy (DPN), familial neuropathies; compression related neuropathy, radicular pain, other infection related neuropathies (eg, leprosy); neuropathy related to: metabolic abnormalities; nutritional factors; vascular insults; inflammation; autoimmune disease; and malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 377 (Actual)
Dates: Start 2010-04; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (63):
- United States (25):
  - Southwest Center for HIV/AIDS, Phoenix, Arizona
  - SW Center for HIV/AIDS, Phoenix, Arizona
  - Arizona Research Center, Phoenix, Arizona
  - AIDS Research Alliance of America, Los Angeles, California
  - Anthony Mills, MD, Inc., Los Angeles, California
  - David Geffen School of Medicine at UCLA c/o NNAB, Los Angeles, California
  - Providence Clinical Research, North Hollywood, California
  - Desert Medical Group, Inc. dba Desert Oasis Healthcare Medical Group, Palm Springs, California
  - University of California San Diego, San Diego, California
  - Stanford University Medical Center, Stanford, California
  - Neuroscience Consultants, LLC., Aventura, Florida
  - South Florida Medical Research, Aventura, Florida
  - The Kinder Medical Group, Miami, Florida
  - Wohlfeiler, Piperato & Associates, LLC, Miami Beach, Florida
  - Meridien Research, Tampa, Florida
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Midtown Neurology, PC, Atlanta, Georgia
  - Neurology Specialists of Decatur Research Center, Decatur, Georgia
  - Rehabilitation Institute of Chicago, Chicago, Illinois
  - Mount Sinai School of Medicine, New York, New York
  - University of Toledo Medical Center, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - University of Texas Physicians, Bellaire, Texas
  - Amelia Court HIV Research Clinic, Dallas, Texas
  - The University of Texas Medical School at Houston, Houston, Texas
- Colombia (4):
  - Asistencia Cientifica de Alta Complejidad, Bogota, Cundinamarca
  - Centro Instituto de Investigaciones Fundación Universitaria Sanitas, Bogota, Cundinamarca
  - Riesgo de Fractura S.A, Bogotá, Cundinamarca
  - Instituto Colombiano para el Avance de la Medicina- Santander S.A.S. - ICAMEDIC Santander S.A.S, Bucaramanga, Santander Department
- Instituto Dominicano de Estudios Virológicos - IDEV, Santo Domingo, Dominican Republic
- India (6):
  - Mahavir Hospital and Research Centre, Hyderabad, Andhra Pradesh
  - Surakshaka Multispeciality Hospital, Hyderabad, Andhra Pradesh
  - Infectious Disease Clinic, Ahmedabad, Gujarat
  - Jaslok Hospital & Research Centre, Mumbai, Maharashtra
  - Deenanath Mangeshkar Hospital and Research Centre, Pune, Maharashtra
  - YR Gaitonde Centre for AIDS Research and Education, Chennai, Tamil Nadu
- Peru (2):
  - Hospital Nacional Dos de Mayo, Lima
  - Hospital Nacional Guillermo Almenara Irigoyen, Lima
- Poland (2):
  - Katedra Chorob Zakaznych i Hepatologii UMK w Toruniu CM w Bydgoszczy, Bydgoszcz
  - Oddzial Diagnostyki i Terapii AIDS, Chorzów
- Puerto Rico (3):
  - Ponce School of Medicine-CAIMED Center, Ponce, PR
  - Ponce School of Medicine - Practice Group, Ponce, PR
  - Puerto Rico Clinical and Translational Research Consortium, Rio Piedras, PR
- South Africa (18):
  - Border Diabetic Centre, East London, Eastern Cape
  - MediSynergy, Port Elizabeth, Eastern Cape
  - Worthwhile Clinical Trials, Benoni, Gauteng
  - Toga Laboratory, Johannesburg, Gauteng
  - Drs Essack and Mitha, Johannesburg, Gauteng
  - University of Witwatersrand-Clinical HIV Research Unit (CHRU), Johannesburg, Gauteng
  - Synexus SA Stanza Bopape Clinical Research Centre, Pretoria, Gauteng
  - Pretoria West Hospital, Pretoria West, Gauteng
  - Chris Hani Baragwanath Hospital, The Palliative Care Centre, Soweto, Gauteng
  - Dr J. Reddy's Surgery, KwaDukuza, KwaZulu-Natal
  - University of Cape Town, Cape Town, Western Cape
  - Synapta Clinical Research Centre, Durban
  - Innovir Institute, Gauteng
  - Mzansi Ethical Research Centre, Middelburg
  - Be Part Yoluntu Centre, Paarl
  - Paarl Research Center, Paarl
  - Clinical Research Unit, University of Pretoria, Pretoria
  - Department of Neurology, Tygerberg
- Thailand (2):
  - South East Asia Research Collaboration with Hawaii, Bangkok
  - Neurology unit, Department of Medicine,, Bangkok

REFERENCES:
- [Derived] Simpson DM, Rice AS, Emir B, Landen J, Semel D, Chew ML, Sporn J. A randomized, double-blind, placebo-controlled trial and open-label extension study to evaluate the efficacy and safety of pregabalin in the treatment of neuropathic pain associated with human immunodeficiency virus neuropathy. Pain. 2014 Oct;155(10):1943-54. doi: 10.1016/j.pain.2014.05.027. Epub 2014 Jun 4. PMID 24907403
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081244&StudyName=Pregabalin%20Versus%20Placebo%20In%20The%20Treatment%20Of%20Neuropathic%20Pain%20Associated%20With%20HIV%20Neuropathy

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants received placebo matched to pregabalin capsule orally twice daily for 2 weeks in placebo lead-in phase prior to randomization.
Groups:
- Pregabalin: Pregabalin 75 milligram (mg) capsule orally twice daily up to Week 1, followed by pregabalin 150 mg capsule orally twice daily up to Week 2, then pregabalin 225 mg capsule orally twice daily up to Week 3, participants who had inadequate pain control and had tolerated pregabalin 225 mg twice daily received pregabalin 300 mg capsule orally twice daily up to Week 4, during 4-week titration (adjustment) phase. Pregabalin capsule 75 mg, 150 mg, 225 mg, or 300 mg orally twice daily (as per tolerability in titration phase) from Week 5 to Week 16, during 12-week maintenance phase. Participants underwent an end-of-study medication taper over a 1-week period.
- Placebo: Placebo matched to pregabalin 75 mg capsule orally twice daily up to Week 1, followed by placebo matched to pregabalin 150 mg capsule orally twice daily up to Week 2, then placebo matched to pregabalin 225 mg capsule orally twice daily up to Week 3, participants who had inadequate pain control and had tolerated placebo matched to pregabalin 225 mg twice daily received placebo matched to pregabalin 300 mg capsule orally twice daily up to Week 4, during 4-week titration (adjustment) phase. Placebo matched to pregabalin capsule 75 mg, 150 mg, 225 mg, or 300 mg orally twice daily (as per tolerability in titration phase) from Week 5 to Week 16, during 12-week maintenance phase. Participants underwent an end-of-study medication taper over a 1-week period.
Period: Overall Study
Arm/Group | Pregabalin | Placebo
Started | 183 | 194
Treated | 183 | 192
Completed | 127 | 131
Not Completed | 56 | 63
Not completed — Adverse Event | 2 | 1
Not completed — Lack of Efficacy | 1 | 1
Not completed — Lost to Follow-up | 3 | 8
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Protocol Violation | 1 | 3
Not completed — Pregnancy | 1 | 0
Not completed — Study Terminated by Sponsor | 43 | 43
Not completed — Other | 1 | 2
Not completed — Randomized but not Treated | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregabalin | Placebo | Total
Number analyzed (Participants) | 183 | 192 | 375
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.2 (9.0) | 42.3 (8.4) | 41.7 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 121 | 116 | 237
  Male | 62 | 76 | 138

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Pain Score at Endpoint (up to Week 16)
Description: Mean pain score was defined as the mean of the last 7 daily diary pain ratings. Participants rated their Human Immunodeficiency Virus (HIV) neuropathy pain over the past 24 hours on an 11-point numeric rating scale ranging from 0 = no pain to 10 = worst possible pain. A rating of 1-3 was considered as mild pain; 4-6 = moderate pain; and 7-10 = severe pain. Endpoint was the last observation for a participant assessed using specified imputation method, modified Baseline Observation Carried Forward (mBOCF).
Time Frame: Baseline, Endpoint (up to Week 16)
Population: Intent to Treat (ITT) population: all randomized participants who took at least 1 dose of study drug. Imputation: mBOCF, baseline data was carried forward for participants who discontinued due to adverse events or had no post-baseline observations; otherwise last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 183 | 192
units on a scale
  Baseline | 6.76 (1.194) | 6.85 (1.222)
  Change at Endpoint | -2.26 (2.200) | -2.36 (2.288)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Analysis of covariance (ANCOVA) model was used with terms of treatment, pooled site, dideoxynucleoside analogue (D-drug) anti-retroviral agent (ART) use and baseline score; Test type: Superiority or Other; p = 0.7090, ANCOVA; Least Squares (LS) Mean Difference = 0.07, 95% CI 2-sided [-0.30 to 0.45], Standard Error of Mean 0.191

2. Secondary Outcome: Number of Participants With Categorical Scores on Patient Global Impression of Change (PGIC)
Description: PGIC: participant rated instrument to measure participant's change in overall status on a 7-point scale; range from 1 (very much improved) to 7 (very much worse). Number of participants in each category is reported.
Time Frame: Week 16
Population: ITT population: all randomized participants who took at least 1 dose of study drug. N (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Number; unit: participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 173 | 176
participants
  Very Much Improved | 42 | 51
  Much Improved | 69 | 66
  Minimally Improved | 42 | 36
  No Change | 13 | 17
  Minimally Worse | 5 | 2
  Much Worse | 2 | 4
  Very Much Worse | 0 | 0
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Overall p-value was derived from Cochran-Mantel-Haenszel (CMH) test adjusted for pooled site and D-drug ART use using modified ridit scores; Test type: Superiority or Other; p = 0.5049, Cochran-Mantel-Haenszel

3. Secondary Outcome: Number of Participants With Categorical Scores on Clinician Global Impression of Change (CGIC)
Description: The CGIC scale measures a physician's global impression of a participant's clinical condition at final visit in terms of change relative to the start of treatment (CGIC). At final visit, the participants CGIC will be categorized into a three point scale as: improvement: CGI response of very much improved, much improved or minimally improved; no change: CGI response of no change; worsening: CGI response of very much worse, much worse or minimally worse. Number of participants in each category is reported.
Time Frame: Week 16
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 172 | 176
participants
  Very Much Improved | 45 | 47
  Much Improved | 59 | 53
  Minimally Improved | 48 | 49
  No Change | 17 | 25
  Minimally Worse | 3 | 2
  Much Worse | 0 | 0
  Very Much Worse | 0 | 0
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.4271, Cochran-Mantel-Haenszel

4. Secondary Outcome: Change From Baseline in Numeric Rating Scale (NRS)-Sleep Interference Score at Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16 and Endpoint (up to Week 16)
Description: Weekly mean sleep interference score was defined as the mean of the daily sleep interference diary ratings split into 7 day intervals. Participants rated how HIV neuropathy pain has interfered with their sleep during the past 24 hours on an 11-point NRS ranging from 0 = does not interfere with sleep to 10 = completely interferes (unable to sleep due to pain). Endpoint was the last observation for a participant assessed using specified imputation method.
Time Frame: Baseline, Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, Endpoint (up to Week 16)
Population: ITT population: all randomized participants who took at least 1 dose of study drug. N (number of participants analyzed) signifies those participants who were evaluable for this measure. n = participants evaluable for this measure at specified time points for each arm group, respectively. Missing data for endpoint (up to Week 16) imputed using LOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 183 | 191
units on a scale
  Baseline (n=183, 191) | 6.55 (1.643) | 6.70 (1.456)
  Change at Week 1 (n=177, 182) | -0.48 (1.067) | -0.37 (1.003)
  Change at Week 2 (n=168, 170) | -0.85 (1.317) | -0.66 (1.292)
  Change at Week 3 (n=163, 163) | -1.09 (1.505) | -0.81 (1.373)
  Change at Week 4 (n=153, 160) | -1.42 (1.804) | -1.20 (1.665)
  Change at Week 5 (n=150, 159) | -1.81 (1.952) | -1.49 (1.824)
  Change at Week 6 (n=144, 152) | -1.95 (2.125) | -1.81 (1.903)
  Change at Week 7 (n=145, 145) | -2.06 (2.234) | -1.94 (1.987)
  Change at Week 8 (n=139, 145) | -2.01 (2.194) | -2.04 (2.103)
  Change at Week 9 (n=135, 137) | -2.45 (2.382) | -2.32 (2.154)
  Change at Week 10 (n=131, 135) | -2.48 (2.315) | -2.39 (2.175)
  Change at Week 11 (n=125, 133) | -2.56 (2.393) | -2.47 (2.207)
  Change at Week 12 (n=122, 131) | -2.69 (2.354) | -2.59 (2.291)
  Change at Week 13 (n=118, 127) | -2.73 (2.337) | -2.82 (2.262)
  Change at Week 14 (n=118, 129) | -2.81 (2.442) | -2.90 (2.346)
  Change at Week 15 (n=117, 127) | -2.90 (2.438) | -2.95 (2.325)
  Change at Week 16 (n=103, 121) | -3.14 (2.475) | -2.94 (2.324)
  Change at Endpoint (n=183, 189) | -2.40 (2.323) | -2.43 (2.296)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Change at Week 1: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.2084, ANCOVA; LS Mean Difference = -0.12, 95% CI 2-sided [-0.31 to 0.07], Standard Error of Mean 0.095
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Change at Week 2: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.1516, ANCOVA; LS Mean Difference = -0.18, 95% CI 2-sided [-0.43 to 0.07], Standard Error of Mean 0.126
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Change at Week 3: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.0468, ANCOVA; LS Mean Difference = -0.28, 95% CI 2-sided [-0.56 to -0.00], Standard Error of Mean 0.142
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Change at Week 4: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.1224, ANCOVA; LS Mean Difference = -0.27, 95% CI 2-sided [-0.62 to 0.07], Standard Error of Mean 0.177
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Change at Week 5: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.0373, ANCOVA; LS Mean Difference = -0.39, 95% CI 2-sided [-0.75 to -0.02], Standard Error of Mean 0.184
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; Change at Week 6: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.1660, ANCOVA; LS Mean Difference = -0.28, 95% CI 2-sided [-0.67 to 0.12], Standard Error of Mean 0.199
Statistical Analysis 7: Comparison: Pregabalin vs Placebo; Change at Week 7: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.3246, ANCOVA; LS Mean Difference = -0.21, 95% CI 2-sided [-0.63 to 0.21], Standard Error of Mean 0.214
Statistical Analysis 8: Comparison: Pregabalin vs Placebo; Change at Week 8: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.4879, ANCOVA; LS Mean Difference = -0.15, 95% CI 2-sided [-0.58 to 0.28], Standard Error of Mean 0.219
Statistical Analysis 9: Comparison: Pregabalin vs Placebo; Change at Week 9: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.2669, ANCOVA; LS Mean Difference = -0.25, 95% CI 2-sided [-0.69 to 0.19], Standard Error of Mean 0.223
Statistical Analysis 10: Comparison: Pregabalin vs Placebo; Change at Week 10: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.5452, ANCOVA; LS Mean Difference = -0.13, 95% CI 2-sided [-0.56 to 0.30], Standard Error of Mean 0.219
Statistical Analysis 11: Comparison: Pregabalin vs Placebo; Change at Week 11: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.5469, ANCOVA; LS Mean Difference = -0.14, 95% CI 2-sided [-0.59 to 0.31], Standard Error of Mean 0.229
Statistical Analysis 12: Comparison: Pregabalin vs Placebo; Change at Week 12: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.7843, ANCOVA; LS Mean Difference = -0.07, 95% CI 2-sided [-0.54 to 0.41], Standard Error of Mean 0.240
Statistical Analysis 13: Comparison: Pregabalin vs Placebo; Change at Week 13: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.9008, ANCOVA; LS Mean Difference = -0.03, 95% CI 2-sided [-0.50 to 0.44], Standard Error of Mean 0.240
Statistical Analysis 14: Comparison: Pregabalin vs Placebo; Change at Week 14: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.9064, ANCOVA; LS Mean Difference = 0.03, 95% CI 2-sided [-0.45 to 0.50], Standard Error of Mean 0.240
Statistical Analysis 15: Comparison: Pregabalin vs Placebo; Change at Week 15: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.7205, ANCOVA; LS Mean Difference = -0.09, 95% CI 2-sided [-0.57 to 0.39], Standard Error of Mean 0.243
Statistical Analysis 16: Comparison: Pregabalin vs Placebo; Change at Week 16: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.4334, ANCOVA; LS Mean Difference = -0.20, 95% CI 2-sided [-0.71 to 0.31], Standard Error of Mean 0.259
Statistical Analysis 17: Comparison: Pregabalin vs Placebo; Change at Endpoint: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.8402, ANCOVA; LS Mean Difference = -0.04, 95% CI 2-sided [-0.43 to 0.35], Standard Error of Mean 0.199

5. Secondary Outcome: Change From Baseline in Numeric Rating Scale (NRS)-Current Pain Score at Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16 and Endpoint (up to Week 16)
Description: Weekly current pain score was defined as the mean of the daily current pain diary ratings split into 7 day intervals. Participants rated current ("right now") HIV neuropathy pain an 11-point NRS ranging from 0 = no pain to 10 = worst possible pain. A rating of 1-3 was considered as mild pain; 4-6 = moderate pain; and 7-10 = severe pain. Endpoint was the last observation for a participant assessed using specified imputation method.
Time Frame: Baseline, Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, Endpoint (up to Week 16)
Population: ITT population: all randomized participants who took at least 1 dose of study drug. n = participants evaluable for this measure at specified time points for each arm group, respectively. Missing data for endpoint (up to Week 16) imputed using LOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 183 | 192
units on a scale
  Baseline (n=183, 192) | 6.66 (1.208) | 6.71 (1.245)
  Change at Week 1 (n=181, 190) | -0.43 (1.000) | -0.34 (0.917)
  Change at Week 2 (n=174, 179) | -0.79 (1.236) | -0.67 (1.282)
  Change at Week 3 (n=170, 172) | -1.10 (1.440) | -0.82 (1.410)
  Change at Week 4 (n=158, 169) | -1.41 (1.682) | -1.17 (1.649)
  Change at Week 5 (n=157, 166) | -1.74 (1.893) | -1.48 (1.845)
  Change at Week 6 (n=152, 157) | -1.87 (2.042) | -1.73 (1.965)
  Change at Week 7 (n=153, 153) | -1.92 (2.074) | -1.88 (2.006)
  Change at Week 8 (n=148, 153) | -2.01 (2.106) | -1.99 (2.105)
  Change at Week 9 (n=143, 148) | -2.30 (2.199) | -2.21 (2.180)
  Change at Week 10 (n=138, 142) | -2.38 (2.172) | -2.24 (2.225)
  Change at Week 11 (n=132, 136) | -2.42 (2.250) | -2.37 (2.218)
  Change at Week 12 (n=128, 135) | -2.55 (2.241) | -2.44 (2.247)
  Change at Week 13 (n=126, 133) | -2.53 (2.241) | -2.60 (2.208)
  Change at Week 14 (n=124, 131) | -2.66 (2.307) | -2.74 (2.303)
  Change at Week 15 (n=120, 132) | -2.77 (2.283) | -2.78 (2.283)
  Change at Week 16 (n=111, 128) | -2.94 (2.370) | -2.81 (2.353)
  Change at Endpoint (n=183, 191) | -2.24 (2.239) | -2.29 (2.302)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Change at Week 1: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.3098, ANCOVA; LS Mean Difference = -0.09, 95% CI 2-sided [-0.25 to 0.08], Standard Error of Mean 0.085
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Change at Week 2: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.2429, ANCOVA; LS Mean Difference = -0.14, 95% CI 2-sided [-0.37 to 0.09], Standard Error of Mean 0.118
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Change at Week 3: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.0504, ANCOVA; LS Mean Difference = -0.27, 95% CI 2-sided [-0.54 to 0.00], Standard Error of Mean 0.137
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Change at Week 4: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.1141, ANCOVA; LS Mean Difference = -0.26, 95% CI 2-sided [-0.58 to 0.06], Standard Error of Mean 0.164
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Change at Week 5: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.0667, ANCOVA; LS Mean Difference = -0.32, 95% CI 2-sided [-0.66 to 0.02], Standard Error of Mean 0.173
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; Change at Week 6: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.2104, ANCOVA; LS Mean Difference = -0.24, 95% CI 2-sided [-0.61 to 0.13], Standard Error of Mean 0.189
Statistical Analysis 7: Comparison: Pregabalin vs Placebo; Change at Week 7: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.4830, ANCOVA; LS Mean Difference = -0.14, 95% CI 2-sided [-0.53 to 0.25], Standard Error of Mean 0.197
Statistical Analysis 8: Comparison: Pregabalin vs Placebo; Change at Week 8: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.5757, ANCOVA; LS Mean Difference = -0.11, 95% CI 2-sided [-0.51 to 0.29], Standard Error of Mean 0.203
Statistical Analysis 9: Comparison: Pregabalin vs Placebo; Change at Week 9: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.3231, ANCOVA; LS Mean Difference = -0.21, 95% CI 2-sided [-0.62 to 0.20], Standard Error of Mean 0.208
Statistical Analysis 10: Comparison: Pregabalin vs Placebo; Change at Week 10: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.3143, ANCOVA; LS Mean Difference = -0.21, 95% CI 2-sided [-0.63 to 0.20], Standard Error of Mean 0.212
Statistical Analysis 11: Comparison: Pregabalin vs Placebo; Change at Week 11: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.6300, ANCOVA; LS Mean Difference = -0.11, 95% CI 2-sided [-0.54 to 0.33], Standard Error of Mean 0.222
Statistical Analysis 12: Comparison: Pregabalin vs Placebo; Change at Week 12: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.5752, ANCOVA; LS Mean Difference = -0.13, 95% CI 2-sided [-0.57 to 0.32], Standard Error of Mean 0.227
Statistical Analysis 13: Comparison: Pregabalin vs Placebo; Change at Week 13: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.8905, ANCOVA; LS Mean Difference = -0.03, 95% CI 2-sided [-0.46 to 0.40], Standard Error of Mean 0.219
Statistical Analysis 14: Comparison: Pregabalin vs Placebo; Change at Week 14: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.9991, ANCOVA; LS Mean Difference = -0.00, 95% CI 2-sided [-0.45 to 0.45], Standard Error of Mean 0.228
Statistical Analysis 15: Comparison: Pregabalin vs Placebo; Change at Week 15: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.8927, ANCOVA; LS Mean Difference = -0.03, 95% CI 2-sided [-0.48 to 0.42], Standard Error of Mean 0.228
Statistical Analysis 16: Comparison: Pregabalin vs Placebo; Change at Week 16: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.8067, ANCOVA; LS Mean Difference = -0.06, 95% CI 2-sided [-0.54 to 0.42], Standard Error of Mean 0.245
Statistical Analysis 17: Comparison: Pregabalin vs Placebo; Change at Endpoint: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.9009, ANCOVA; LS Mean Difference = 0.02, 95% CI 2-sided [-0.35 to 0.40], Standard Error of Mean 0.190

6. Secondary Outcome: Change From Baseline in Brief Pain Inventory-Short Form (BPI-sf) Score at Week 4, 8, 12, 16 and Endpoint (up to Week 16)
Description: BPI-sf:5-item self-administered questionnaire to assess severity,impact of pain on daily functions. Pain Severity Index (PSI):average of Question 1-4 each measured severity of pain over past 24-hours on 11-point scale (0=no pain to 10=worst possible pain). Pain Interference Index (PII):average of 7 pain interference items of Question 5 that measured level of interference of pain on daily function on 11-point scale (0=does not interfere to 10=completely interferes). For PSI, PII range:0-10 higher score=higher pain/interference. Endpoint=last observation for participant as per imputation method.
Time Frame: Baseline, Week 4, 8, 12, 16, Endpoint (up to Week 16)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 182 | 192
units on a scale
  Baseline: PSI (n=182, 192) | 6.49 (1.175) | 6.47 (1.292)
  Change at Week 4: PSI (n=158, 169) | -1.55 (1.725) | -1.28 (1.811)
  Change at Week 8: PSI (n=146, 154) | -2.15 (2.142) | -2.02 (2.117)
  Change at Week 12: PSI (n=126, 137) | -2.49 (2.311) | -2.60 (2.169)
  Change at Week 16: PSI (n=166, 166) | -2.38 (2.335) | -2.55 (2.354)
  Change at Endpoint: PSI (n=175,182) | -2.36 (2.291) | -2.44 (2.334)
  Baseline: PII (n=182, 192) | 5.51 (1.963) | 5.44 (2.013)
  Change at Week 4: PII (n=158, 169) | -1.43 (2.068) | -1.40 (2.358)
  Change at Week 8: PII (n=146, 154) | -2.00 (2.319) | -1.97 (2.312)
  Change at Week 12: PII (n=126, 137) | -2.32 (2.450) | -2.32 (2.183)
  Change at Week 16: PII (n=166, 165) | -2.14 (2.434) | -2.38 (2.290)
  Change at Endpoint: PII (n=175,182) | -2.12 (2.415) | -2.31 (2.306)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Change at Week 4, PSI: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.0948, ANCOVA; LS Mean Difference = -0.30, 95% CI 2-sided [-0.64 to 0.05], Standard Error of Mean 0.177
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Change at Week 8, PSI: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.4167, ANCOVA; LS Mean Difference = -0.17, 95% CI 2-sided [-0.57 to 0.23], Standard Error of Mean 0.203
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Change at Week 12, PSI: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.8179, ANCOVA; LS Mean Difference = 0.05, 95% CI 2-sided [-0.39 to 0.50], Standard Error of Mean 0.226
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Change at Week 16, PSI: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.6913, ANCOVA; LS Mean Difference = 0.08, 95% CI 2-sided [-0.33 to 0.50], Standard Error of Mean 0.209
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Change at Endpoint, PSI: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.9475, ANCOVA; LS Mean Difference = 0.01, 95% CI 2-sided [-0.39 to 0.41], Standard Error of Mean 0.203
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; Change at Week 4, PII: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.7412, ANCOVA; LS Mean Difference = -0.07, 95% CI 2-sided [-0.47 to 0.33], Standard Error of Mean 0.204
Statistical Analysis 7: Comparison: Pregabalin vs Placebo; Change at Week 8, PII: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.9715, ANCOVA; LS Mean Difference = 0.01, 95% CI 2-sided [-0.41 to 0.43], Standard Error of Mean 0.213
Statistical Analysis 8: Comparison: Pregabalin vs Placebo; Change at Week 12, PII: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.8163, ANCOVA; LS Mean Difference = 0.05, 95% CI 2-sided [-0.38 to 0.48], Standard Error of Mean 0.218
Statistical Analysis 9: Comparison: Pregabalin vs Placebo; Change at Week 16, PII: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.3682, ANCOVA; LS Mean Difference = 0.18, 95% CI 2-sided [-0.22 to 0.58], Standard Error of Mean 0.204
Statistical Analysis 10: Comparison: Pregabalin vs Placebo; Change at Endpoint, PII: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.3511, ANCOVA; LS Mean Difference = 0.19, 95% CI 2-sided [-0.21 to 0.58], Standard Error of Mean 0.199

7. Secondary Outcome: Change From Baseline in Neuropathic Pain Symptom Inventory (NPSI) Item Scores at Endpoint (up to Week 16)
Description: NPSI: participant-rated questionnaire to evaluate different symptoms of neuropathic pain. It includes 10 descriptors and 2 temporal items. Results reported for the 10 descriptors (burning, squeezing, pressure, electric shocks, stabbing, light touching of area, pressure of area, cold of area, pins and needles, tingling) quantified on a 0 (no symptoms) to 10 (worst symptoms imaginable) scale. Endpoint was the last observation for a participant assessed using specified imputation method.
Time Frame: Baseline, Endpoint (up to Week 16)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 183 | 192
units on a scale
  Baseline: Burning (n=183, 192) | 6.1 (2.33) | 6.2 (2.52)
  Change at Endpoint: Burning (n=173, 176) | -2.4 (2.91) | -2.6 (3.06)
  Baseline: Squeezing (n=183, 192) | 5.3 (2.57) | 5.2 (2.98)
  Change at Endpoint: Squeezing (n=173, 176) | -2.1 (3.02) | -2.1 (3.03)
  Baseline: Pressure (n=183, 192) | 5.8 (2.50) | 5.5 (2.73)
  Change at Endpoint: Pressure (n=172, 176) | -2.3 (3.19) | -2.2 (3.15)
  Baseline: Electric Shocks (n=183, 192) | 5.4 (2.76) | 5.1 (2.84)
  Change at Endpoint: Electric Shocks (n=173, 176) | -2.2 (3.18) | -2.0 (3.10)
  Baseline: Stabbing (n=183, 192) | 5.8 (2.46) | 6.1 (2.58)
  Change at Endpoint: Stabbing (n=173, 176) | -2.2 (3.00) | -2.5 (3.11)
  Baseline: Light Touching (n=183, 192) | 5.0 (2.60) | 5.0 (2.62)
  Change at Endpoint: Light Touching (n=173, 176) | -1.9 (2.91) | -1.9 (3.05)
  Baseline: Pressure of Area (n=183, 192) | 6.0 (2.12) | 6.0 (2.25)
  Change at Endpoint: Pressure of Area (n=173, 176) | -2.5 (2.75) | -2.3 (2.99)
  Baseline: Cold of Area (n=183, 192) | 5.9 (2.56) | 5.5 (2.87)
  Change at Endpoint: Cold of Area (n=173, 176) | -2.2 (2.98) | -2.0 (3.07)
  Baseline: Pins and Needles (n=183, 192) | 6.7 (2.14) | 6.6 (2.23)
  Change at Endpoint: Pins and Needles (n=173, 176) | -2.6 (2.90) | -2.6 (3.12)
  Baseline: Tingling (n=183, 192) | 5.8 (2.49) | 6.1 (2.42)
  Change at Endpoint: Tingling (n=173, 176) | -2.1 (3.01) | -2.4 (3.09)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Change at Endpoint, Burning: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.9686, ANCOVA; LS Mean Difference = 0.0, 95% CI 2-sided [-0.5 to 0.5], Standard Error of Mean 0.25
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Change at Endpoint, Squeezing: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.4476, ANCOVA; LS Mean Difference = -0.2, 95% CI 2-sided [-0.6 to 0.3], Standard Error of Mean 0.23
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Change at Endpoint, Pressure: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.5630, ANCOVA; LS Mean Difference = -0.1, 95% CI 2-sided [-0.6 to 0.3], Standard Error of Mean 0.24
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Change at Endpoint, Electric Shocks: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.9937, ANCOVA; LS Mean Difference = 0.0, 95% CI 2-sided [-0.5 to 0.5], Standard Error of Mean 0.25
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Change at Endpoint, Stabbing: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.8718, ANCOVA; LS Mean Difference = 0.0, 95% CI 2-sided [-0.5 to 0.5], Standard Error of Mean 0.25
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; Change at Endpoint, Light Touching: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.8241, ANCOVA; LS Mean Difference = -0.1, 95% CI 2-sided [-0.5 to 0.4], Standard Error of Mean 0.24
Statistical Analysis 7: Comparison: Pregabalin vs Placebo; Change at Endpoint, Pressure of Area: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.3164, ANCOVA; LS Mean Difference = -0.2, 95% CI 2-sided [-0.7 to 0.2], Standard Error of Mean 0.25
Statistical Analysis 8: Comparison: Pregabalin vs Placebo; Change at Endpoint, Cold of Area: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.8996, ANCOVA; LS Mean Difference = -0.0, 95% CI 2-sided [-0.5 to 0.5], Standard Error of Mean 0.25
Statistical Analysis 9: Comparison: Pregabalin vs Placebo; Change at Endpoint, Pins and Needles: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.9676, ANCOVA; LS Mean Difference = -0.0, 95% CI 2-sided [-0.5 to 0.5], Standard Error of Mean 0.26
Statistical Analysis 10: Comparison: Pregabalin vs Placebo; Change at Endpoint, Tingling: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.9091, ANCOVA; LS Mean Difference = -0.0, 95% CI 2-sided [-0.5 to 0.5], Standard Error of Mean 0.25

8. Secondary Outcome: Neuropathic Pain Symptom Inventory (NPSI): Change From Baseline in Number of Participants With Duration of Spontaneous Pain and Number of Pain Attacks at Endpoint (up to Week 16)
Description: NPSI: participant-rated questionnaire to evaluate different symptoms of neuropathic pain. It includes 10 descriptors, and 2 temporal items. Results reported for categorical change in temporal items assessed on 5-point scale for duration of spontaneous pain (1=continuously, 2=8-12 hours [hrs], 3=4-7 hrs, 4=1-3 hrs, 5=less than 1 hr), numbers of pain attacks (1=more than 20, 2=11-20 attacks, 3=6-10 attacks, 4=1-5 attacks, 5=no attack). Change data categorized as worsened (negative change), unchanged (no change), and improved (positive change). Endpoint=last observation as per imputation method.
Time Frame: Baseline, Endpoint (up to Week 16)
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 173 | 176
participants
  Duration of Spontaneous Pain, Worsened (n=173,172) | 31 | 33
  Duration of Spontaneous Pain, Unchanged(n=173,172) | 56 | 50
  Duration of Spontaneous Pain, Improved (n=173,172) | 86 | 89
  Number of Pain Attacks, Worsened (n=173, 176) | 40 | 25
  Number of Pain Attacks, Unchanged (n=173, 176) | 49 | 54
  Number of Pain Attacks, Improved (n=173, 176) | 84 | 97
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Duration of Spontaneous Pain: Overall p-value was derived from CMH test adjusted for pooled site and D-drug ART use using modified ridit scores; Test type: Superiority or Other; p = 0.7300, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Number of Pain Attacks: Overall p-value was derived from CMH test adjusted for pooled site and D-drug ART use using modified ridit scores; Test type: Superiority or Other; p = 0.0559, Cochran-Mantel-Haenszel

9. Secondary Outcome: Change From Baseline in Neuropathic Pain Symptom Inventory (NPSI) Subscales and Total Intensity Score at Endpoint (up to Week 16)
Description: NPSI: participant rated questionnaire to evaluate different symptoms of neuropathic pain (subscales: burning [superficial] spontaneous pain, pressing [deep] spontaneous pain, paroxysmal pain, evoked pain, and paresthesia/dyesthesia [P/D]). Includes 10 descriptors quantified on a 0 (no symptoms) to 10 (worst symptoms imaginable) and 2 temporal items assessing duration of spontaneous ongoing and paroxysmal pain. The relevant subscales and total score were transformed to 0-1, higher score indicates a greater intensity of pain. Endpoint=last observation for participant as per imputation method.
Time Frame: Baseline, Endpoint (up to Week 16)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 183 | 192
units on a scale
  Baseline: Burning Pain (n=183, 192) | 0.61 (0.233) | 0.62 (0.252)
  Change at Endpoint: Burning Pain (n=173, 176) | -0.24 (0.291) | -0.26 (0.306)
  Baseline: Pressing Pain (n=182, 192) | 0.55 (0.227) | 0.54 (0.248)
  Change at Endpoint: Pressing Pain (n=173, 176) | -0.22 (0.280) | -0.21 (0.279)
  Baseline: Paroxysmal Pain (n=183, 192) | 0.56 (0.227) | 0.56 (0.236)
  Change at Endpoint: Paroxysmal Pain (n=173, 176) | -0.22 (0.272) | -0.23 (0.279)
  Baseline: Evoked Pain (n=183, 192) | 0.57 (0.202) | 0.55 (0.206)
  Change at Endpoint: Evoked Pain (n=173, 176) | -0.22 (0.243) | -0.21 (0.253)
  Baseline: P/D (n=183, 192) | 0.62 (0.211) | 0.63 (0.199)
  Change at Endpoint: P/D (n=173, 176) | -0.23 (0.282) | -0.25 (0.277)
  Baseline: Total Score (n=182, 192) | 0.58 (0.173) | 0.57 (0.175)
  Change at Endpoint: Total Score (n=173,176) | -0.22 (0.231) | -0.23 (0.236)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Change at Endpoint, Burning Pain: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.9686, ANCOVA; LS Mean Difference = 0.00, 95% CI 2-sided [-0.05 to 0.05], Standard Error of Mean 0.025
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Change at Endpoint, Pressing Pain: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.4711, ANCOVA; LS Mean Difference = -0.02, 95% CI 2-sided [-0.06 to 0.03], Standard Error of Mean 0.022
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Change at Endpoint, Paroxysmal Pain: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.9215, ANCOVA; LS Mean Difference = 0.00, 95% CI 2-sided [-0.04 to 0.05], Standard Error of Mean 0.023
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Change at Endpoint, Evoked Pain: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.6042, ANCOVA; LS Mean Difference = -0.01, 95% CI 2-sided [-0.05 to 0.03], Standard Error of Mean 0.021
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Change at Endpoint, P/D: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.9394, ANCOVA; LS Mean Difference = -0.00, 95% CI 2-sided [-0.05 to 0.04], Standard Error of Mean 0.024
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; Change at Endpoint, Total Score: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.7801, ANCOVA; LS Mean Difference = -0.01, 95% CI 2-sided [-0.04 to 0.03], Standard Error of Mean 0.020

10. Secondary Outcome: Total Sleep Time (TST) and Minutes of Interrupted Sleep (MIS)
Description: Total sleep time is the number of minutes asleep between time of sleep onset to morning awakening and MIS is the number of minutes spent awake after sleep onset to final awakening. TST and MIS were determined by actigraphy. Actigraphy was performed with an accelerometer that was worn on the wrist like a watch. It was programmed to record movements while the device was being worn. Endpoint was the last observation for a participant assessed using specified imputation method.
Time Frame: Baseline (Day -14 to 1), Week 1 through Week 4, Week 12 through Week 16, Endpoint (up to Week 16)
Population: ITT population. N (number of participants analyzed) = participants evaluable for this measure. Missing data for endpoint (up to Week 16) imputed using LOCF. Data for Baseline (Day -14 to 1), Week 1 through Week 4, Week 12 through Week 16 were collected and reported in individual participant listings but not statistically summarized for analysis.
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 155 | 152
minutes
  Endpoint: TST | 396.84 (5.04) | 400.29 (5.29)
  Endpoint: MIS | 41.48 (1.45) | 45.14 (1.50)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Endpoint TST: ANCOVA model was used with treatment as a fixed effect and D-drug ART, pooled site value, baseline value as covariates; Test type: Superiority or Other; p = 0.6012, ANCOVA; LS Mean Difference = -3.44, Standard Error of Mean 6.58
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Endpoint MIS: ANCOVA model was used with treatment as a fixed effect and D-drug ART, pooled site value, baseline value as covariates; Test type: Superiority or Other; p = 0.0534, ANCOVA; LS Mean Difference = -3.66, Standard Error of Mean 1.89

11. Secondary Outcome: Sleep Fragmentation Index (SFI)
Description: SFI is a measure to quantify sleep restlessness. SFI calculated from analysis of the periods that participant was not moving (immobile bouts). It is number of immobile bouts that were exactly 1 minute long divided by total number of immobile bouts. Value ranges from 0-100 percent, with low number representing more restful sleep. SFI determined by actigraphy. Actigraphy was performed with an accelerometer that was worn on wrist like a watch. It was programmed to record movements while device was being worn. Endpoint was the last observation for a participant assessed using imputation method.
Time Frame: Baseline (Day -14 to 1), Week 1 through Week 4, Week 12 through Week 16, Endpoint (up to Week 16)
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: percentage of immobile bouts
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 155 | 151
percentage of immobile bouts | 18.57 (0.47) | 19.60 (0.49)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; ANCOVA model was used with treatment as a fixed effect and D-drug ART, pooled site value, baseline value as covariates; Test type: Superiority or Other; p = 0.0966, ANCOVA; LS Mean Difference = -1.03, Standard Error of Mean 0.62

12. Secondary Outcome: Sleep Efficiency
Description: Sleep efficiency is the time spent asleep divided by total time between sleep onset and sleep end, multiplied by 100. Sleep efficiency was determined by actigraphy. Actigraphy was performed with an accelerometer that was worn on the wrist like a watch. It was programmed to record movements while the device was being worn. Endpoint was the last observation for a participant assessed using specified imputation method.
Time Frame: Baseline (Day -14 to 1), Week 1 through Week 4, Week 12 through Week 16, Endpoint (up to Week 16)
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: Percent time between sleep onset and end
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 155 | 151
Percent time between sleep onset and end | 85.80 (0.39) | 84.84 (0.41)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; ANCOVA model was used with treatment as a fixed effect and D-drug ART, pooled site value, baseline value as covariates; Test type: Superiority or Other; p = 0.0611, ANCOVA; LS Mean Difference = 0.97, Standard Error of Mean 0.51

13. Secondary Outcome: Total Activity Counts
Description: Activity counts are the units of motion. It is equal to the sum of peak accelerations each second during the epoch (60 seconds). Total activity counts per day is the sum of the activity counts for each epoch (60 seconds) during the "day" (non sleep period). A total activity count was determined by actigraphy. Actigraphy was performed with an accelerometer that was worn on the wrist like a watch. It was programmed to record movements while the device was being worn. Endpoint was the last observation for a participant assessed using specified imputation method.
Time Frame: Baseline (Day -14 to 1), Week 1 through Week 4, Week 12 through Week 16, Endpoint (up to Week 16)
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: activity counts per day
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 152 | 151
activity counts per day | 297350 (5280.2) | 305787 (5480.9)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; ANCOVA model was used with treatment as a fixed effect and D-drug ART, pooled site value, baseline value as covariates; Test type: Superiority or Other; p = 0.2195, ANCOVA; LS Mean Difference = -8436, Standard Error of Mean 6855.2

14. Secondary Outcome: Percentage Day Time Above Sedentary Level
Description: Percentage of time above sedentary level is number of epochs (60 seconds) with greater than (>) 200 activity counts per minute divided by total number of epochs during the "day" (non sleep period) multiplied by 100. This was determined by actigraphy. Actigraphy was performed with an accelerometer that was worn on the wrist like a watch. It was programmed to record movements while the device was being worn. Endpoint was the last observation for a participant assessed using specified imputation method.
Time Frame: Baseline (Day -14 to 1), Week 1 through Week 4, Week 12 through Week 16, Endpoint (up to Week 16)
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: percentage of day time
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 155 | 152
percentage of day time | 52.43 (0.51) | 52.28 (0.53)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Non-Inferiority or Equivalence — ANCOVA model was used with treatment as a fixed effect and D-drug ART, pooled site value, baseline value as covariates; p = 0.8241, ANCOVA; LS Mean Difference = 0.15, Standard Error of Mean 0.66

15. Secondary Outcome: Change From Baseline in Medical Outcomes Study-Sleep Scale (MOS-SS) at Endpoint (up to Week 16)
Description: Participant-rated 12-item questionnaire to assess constructs of sleep over past week; 7 subscales: sleep disturbance (range 0-100), snoring (range 0-100), awaken short of breath (SOB) or with headache (range 0-100), sleep adequacy (range 0-100), somnolence (range: 0-100); sleep quantity (range: 0-24), optimal sleep (yes/no), and 9 item index measures of sleep disturbance provide composite scores: sleep problems index (range 0-100). Except adequacy, optimal sleep and quantity, higher scores=more impairment. Endpoint was the last observation for a participant assessed using imputation method.
Time Frame: Baseline, Endpoint (up to Week 16)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 183 | 192
units on a scale
  Baseline: Sleep Disturbance (n=183, 192) | 35.27 (22.127) | 39.32 (22.800)
  Change at Endpoint: Sleep Disturbance (n=173, 175) | -6.58 (22.856) | -8.64 (25.317)
  Baseline: Snoring (n=181, 192) | 25.30 (31.456) | 26.04 (34.077)
  Change at Endpoint: Snoring (n=171, 175) | 0.94 (35.301) | -3.77 (33.862)
  Baseline: SOB (n= 183, 192) | 22.08 (27.216) | 25.83 (28.567)
  Change at Endpoint: SOB (n=173, 175) | -3.01 (28.938) | -7.09 (30.552)
  Baseline: Quantity (n= 183, 192) | 7.50 (1.969) | 7.96 (3.976)
  Change at Endpoint: Quantity (n=173, 175) | 0.27 (1.814) | 0.36 (2.082)
  Baseline: Adequacy (n= 183, 192) | 57.81 (25.776) | 54.22 (24.801)
  Change at Endpoint: Adequacy (n=173, 175) | 5.26 (30.319) | 4.63 (30.091)
  Baseline: Somnolence (n= 183, 192) | 26.05 (21.078) | 29.10 (20.773)
  Change at Endpoint: Somnolence (n=173, 175) | -0.77 (22.946) | -4.23 (24.136)
  Baseline: Sleep Problems Index (n= 183, 192) | 32.97 (16.726) | 36.91 (16.862)
  Change at Endpoint:Sleep Problems Index(n=173,175) | -4.25 (17.382) | -6.70 (18.358)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Change at Endpoint, Sleep Disturbance: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.8528, ANCOVA; LS Mean Difference = -0.38, 95% CI 2-sided [-4.42 to 3.66], Standard Error of Mean 2.052
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Change at Endpoint, Snoring: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.3650, ANCOVA; LS Mean Difference = 2.88, 95% CI 2-sided [-3.37 to 9.14], Standard Error of Mean 3.179
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Change at Endpoint, SOB: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.7237, ANCOVA; LS Mean Difference = 0.89, 95% CI 2-sided [-4.07 to 5.86], Standard Error of Mean 2.525
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Change at Endpoint, Quantity: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.2783, ANCOVA; LS Mean Difference = -0.18, 95% CI 2-sided [-0.50 to 0.15], Standard Error of Mean 0.165
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Change at Endpoint, Adequacy: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.2475, ANCOVA; LS Mean Difference = 3.02, 95% CI 2-sided [-2.11 to 8.16], Standard Error of Mean 2.611
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; Change at Endpoint, Somnolence: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.5492, ANCOVA; LS Mean Difference = 1.16, 95% CI 2-sided [-2.64 to 4.96], Standard Error of Mean 1.933
Statistical Analysis 7: Comparison: Pregabalin vs Placebo; Change at Endpoint, Sleep Problems Index: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.9113, ANCOVA; LS Mean Difference = 0.18, 95% CI 2-sided [-3.00 to 3.36], Standard Error of Mean 1.614

16. Secondary Outcome: Medical Outcomes Study-Sleep Scale (MOS-SS): Number of Participants With Optimal Sleep
Description: MOS-SS: participant-rated 12 item questionnaire to assess constructs of sleep over past week. It included 7 subscales: sleep disturbance, snoring, awaken short of breath or with headache, sleep adequacy, somnolence, sleep quantity, optimal sleep, and 9 item index measures of sleep disturbance provide composite scores: sleep problems index. Participants responded whether their sleep was optimal or not optimal by choosing yes or no. Endpoint was the last observation for a participant assessed using imputation method.
Time Frame: Baseline, Endpoint (up to Week 16)
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 183 | 192
participants
  Baseline (n=183, 192) | 80 | 77
  Endpoint (n=173, 176) | 80 | 80
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Endpoint: Overall p-value was derived from CMH test adjusted for pooled site and D-drug ART use using modified ridit scores; Test type: Superiority or Other; p = 0.7399, Cochran-Mantel-Haenszel

17. Secondary Outcome: Change From Baseline in Hospital Anxiety and Depression Scales (HADS) at Endpoint (up to Week 16)
Description: HADS: participant rated questionnaire with 2 subscales. HADS-A assesses state of generalized anxiety (anxious mood, restlessness, anxious thoughts, panic attacks); HADS-D assesses state of lost interest and diminished pleasure response (lowering of hedonic tone). Each subscale comprised of 7 items with range 0 (no presence of anxiety or depression) to 3 (severe feeling of anxiety or depression). Total score 0 to 21 for each subscale; higher score indicates greater severity of anxiety and depression symptoms. Endpoint was the last observation for a participant assessed using imputation method.
Time Frame: Baseline, Endpoint (up to Week 16)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 183 | 192
units on a scale
  Baseline: HADS-A (n=183, 192) | 5.99 (4.065) | 6.32 (4.216)
  Change at Endpoint: HADS-A (n=173, 176) | -1.03 (4.550) | -1.50 (4.593)
  Baseline: HADS-D (n=183, 192) | 4.92 (3.478) | 5.42 (3.885)
  Change at Endpoint: HADS-D (n=173, 176) | 0.07 (4.238) | -1.02 (4.038)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Change at Endpoint, HADS-A: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.8258, ANCOVA; LS Mean Difference = 0.08, 95% CI 2-sided [-0.67 to 0.84], Standard Error of Mean 0.386
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Change at Endpoint, HADS-D: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.0840, ANCOVA; LS Mean Difference = 0.65, 95% CI 2-sided [-0.09 to 1.38], Standard Error of Mean 0.372

18. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) at Endpoint (up to Week 16)
Description: SF-36 is a standardized survey evaluating 8 domains of functional health and well being: physical and social (So) functioning (Fn), physical and emotional role (role-physical [R-P], role-emotional [R-E]) limitations, bodily pain (BP), general health (GH), vitality (Vit), mental health (MnH). Two summary scores include Physical Component (Ph C) and Mental Component (Mn C). The score for a section is an average of the individual question scores. Score range for domain scores and summary scores: 0-100 (100=highest level of functioning).
Time Frame: Baseline, Endpoint (up to Week 16)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 183 | 192
units on a scale
  Baseline: Ph Fn (n=183, 192) | 55.25 (24.913) | 56.30 (24.444)
  Change at Endpoint: Ph Fn (n=173, 176) | 8.29 (26.438) | 6.85 (27.839)
  Baseline: R-P (n=183, 192) | 55.43 (25.806) | 58.37 (25.078)
  Change at Endpoint: R-P (n=173, 176) | 9.03 (27.012) | 7.05 (29.122)
  Baseline: BP (n=183, 192) | 48.11 (20.149) | 48.47 (21.855)
  Change at Endpoint: BP (n=172, 176) | 13.13 (24.846) | 12.86 (28.888)
  Baseline: GH (n=183, 192) | 58.83 (20.583) | 59.47 (19.808)
  Change at Endpoint: GH (n=173, 176) | 8.25 (20.985) | 7.37 (21.300)
  Baseline: Ph C (n=183, 192) | 39.66 (8.632) | 40.06 (8.110)
  Change at Endpoint: Ph C (n=171, 176) | 4.44 (8.530) | 4.17 (9.528)
  Baseline: Vit (n=183, 192) | 61.01 (16.338) | 59.80 (18.443)
  Change at Endpoint: Vit (n=172, 176) | 2.86 (19.196) | 4.87 (21.014)
  Baseline: So Fn (n=183, 192) | 68.37 (22.498) | 66.34 (22.825)
  Change at Endpoint: So Fn (n=173, 176) | 2.60 (26.866) | 6.18 (23.299)
  Baseline: R-E (n=183, 192) | 63.80 (26.333) | 67.93 (25.214)
  Change at Endpoint: R-E (n=173, 176) | 6.74 (29.536) | 1.85 (29.307)
  Baseline: MnH (n=183, 192) | 69.07 (16.902) | 68.59 (19.133)
  Change at Endpoint: MnH (n=172, 176) | 3.11 (20.698) | 4.12 (19.776)
  Baseline: Mn C (n=183, 192) | 47.12 (10.037) | 47.18 (10.473)
  Change at Endpoint: Mn C (n=171, 176) | 1.18 (11.394) | 1.21 (10.519)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Change at Endpoint, Ph Fn: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.6114, ANCOVA; LS Mean Difference = 1.22, 95% CI 2-sided [-3.49 to 5.92], Standard Error of Mean 2.393
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Change at Endpoint, R-P: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.8209, ANCOVA; LS Mean Difference = 0.57, 95% CI 2-sided [-4.39 to 5.53], Standard Error of Mean 2.522
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Change at Endpoint, BP: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.9737, ANCOVA; LS Mean Difference = 0.08, 95% CI 2-sided [-4.52 to 4.67], Standard Error of Mean 2.335
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Change at Endpoint, GH: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.6966, ANCOVA; LS Mean Difference = 0.76, 95% CI 2-sided [-3.05 to 4.57], Standard Error of Mean 1.937
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Change at Endpoint, Ph C: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.8569, ANCOVA; LS Mean Difference = 0.15, 95% CI 2-sided [-1.44 to 1.73], Standard Error of Mean 0.807
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; Change at Endpoint, Vit: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.4734, ANCOVA; LS Mean Difference = -1.33, 95% CI 2-sided [-4.96 to 2.31], Standard Error of Mean 1.847
Statistical Analysis 7: Comparison: Pregabalin vs Placebo; Change at Endpoint, So Fn: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.3625, ANCOVA; LS Mean Difference = -1.97, 95% CI 2-sided [-6.22 to 2.28], Standard Error of Mean 2.159
Statistical Analysis 8: Comparison: Pregabalin vs Placebo; Change at Endpoint, R-E: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.2736, ANCOVA; LS Mean Difference = 2.79, 95% CI 2-sided [-2.21 to 7.79], Standard Error of Mean 2.543
Statistical Analysis 9: Comparison: Pregabalin vs Placebo; Change at Endpoint, MnH: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.8199, ANCOVA; LS Mean Difference = -0.41, 95% CI 2-sided [-3.98 to 3.15], Standard Error of Mean 1.811
Statistical Analysis 10: Comparison: Pregabalin vs Placebo; Change at Endpoint, Mn C: ANCOVA model was used with terms of treatment, pooled site, D-drug ART use and baseline score; Test type: Superiority or Other; p = 0.9361, ANCOVA; LS Mean Difference = 0.08, 95% CI 2-sided [-1.82 to 1.98], Standard Error of Mean 0.967

19. Secondary Outcome: Number of Participants Who Were Employed or Unemployed Assessed by Work Productivity and Activity Impairment: Specific Health Problem (WPAI: SHP) Questionnaire
Description: WPAI: 6-question participant rated questionnaire to determine the degree to which specific health problem (SHP) affected work productivity while at work and affected activities outside of work. It assesses amount of absenteeism, presenteeism and daily activity impairment attributable to a HIV neuropathy pain. Number of participants who responded "Yes/No" to Question 1: Are you currently employed (working for pay)? are reported.
Time Frame: Baseline, Week 16, 17
Population: ITT population: all randomized participants who took at least 1 dose of study drug. n = participants evaluable for this measure at specified time points for each arm group, respectively.
Measure: Number; unit: participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 183 | 192
participants
  Baseline: Employed (n=183, 192) | 57 | 57
  Week 16: Employed (n=169, 170) | 57 | 51
  Week 17: Employed (n=167, 171) | 58 | 47
  Baseline: Unemployed (n=183, 192) | 126 | 135
  Week 16: Unemployed (n=169, 170) | 112 | 119
  Week 17: Unemployed (n=167, 171) | 109 | 124

20. Secondary Outcome: Absenteeism and Presenteeism Assessed by Work Productivity and Activity Impairment: Specific Health Problem (WPAI: SHP) Questionnaire
Description: WPAI: 6-question participant rated questionnaire to determine the degree to which SHP affected work productivity while at work and affected activities outside of work. It assesses amount of absenteeism, presenteeism and daily activity impairment attributable to a HIV neuropathy pain. Question 2 and 3 assesses absenteeism as: Hours of work missed in past 7 days due to leg/foot pain or other reason, respectively. Question 4 assesses presenteeism as: Hours of work performed in past 7 days. A participant who had responded 'no' to question 1 regarding employment status reported hours of work and as this was a self-reported questionnaire the source data were included.
Time Frame: Baseline, Week 16, 17
Population: ITT population: all randomized participants who took at least 1 dose of study drug. N (number of participants analyzed) signifies those participants who were evaluable for this measure. n = participants evaluable for this measure at specified time points for each arm group, respectively.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 58 | 58
hours
  Baseline, Hours Missed,Leg/Foot Pain (n=57, 58) | 5.58 (10.601) | 4.86 (11.488)
  Week 16, Hours Missed,Leg/Foot Pain (n=57, 54) | 2.05 (5.044) | 2.41 (6.603)
  Week 17, Hours Missed,Leg/Foot Pain (n=58, 48) | 3.03 (5.364) | 1.27 (2.703)
  Baseline, Hours Missed,Other Reason (n=57, 58) | 12.77 (21.253) | 7.31 (15.144)
  Week 16, Hours Missed,Other Reason (n=57, 54) | 7.53 (15.121) | 6.74 (14.070)
  Week 17, Hours Missed,Other Reason (n=58, 48) | 7.72 (17.887) | 2.94 (6.635)
  Baseline: Hours Worked (n=57, 58) | 32.54 (17.367) | 28.76 (18.780)
  Week 16: Hours Worked (n=57, 54) | 37.44 (19.441) | 32.72 (19.835)
  Week 17: Hours Worked (n=58, 48) | 34.83 (20.670) | 38.15 (21.399)

21. Secondary Outcome: Productivity and Activity Impairment Assessed by Work Productivity and Activity Impairment: Specific Health Problem (WPAI: SHP) Questionnaire
Description: WPAI: 6-question participant rated questionnaire to determine the degree to which SHP affected work productivity while at work and affected activities outside of work. It assesses amount of absenteeism, presenteeism and daily activity impairment attributable to a HIV neuropathy pain. Question 5 and 6 assesses: How much leg/foot pain affect productivity and daily activity, respectively in past 7 days? on 11-point scale, where 0 (not affected/no impairment) to 10 (completely affected/impaired).
Time Frame: Baseline, Week 16, 17
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 183 | 192
units on a scale
  Baseline: Productivity Affected (n=55, 57) | 5.00 (2.480) | 5.93 (2.513)
  Week 16: Productivity Affected (n=60, 54) | 3.60 (2.402) | 3.15 (2.771)
  Week 17: Productivity Affected (n=58, 48) | 3.40 (2.615) | 3.00 (2.806)
  Baseline: Daily Activity Affected (n=183, 192) | 6.03 (2.078) | 6.12 (2.190)
  Week 16: Daily Activity Affected (n=169, 170) | 3.75 (2.547) | 3.66 (2.769)
  Week 17: Daily Activity Affected (n=167, 171) | 3.82 (2.568) | 3.64 (2.754)

22. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent (TE) Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Baseline up to 28 days after last dose
Population: Safety population included all participants who signed the informed consent, had exposure to study drug and had at least one safety assessment.
Measure: Number; unit: participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 183 | 192
participants
  AEs | 126 | 117
  SAEs | 7 | 7

23. Other Pre Specified Outcome: Number of Participants With Abnormal Laboratory Test Findings
Description: Laboratory tests included hematology, chemistry, cluster of differentiation 4 (CD4) count and cluster of differentiation 8 (CD8) count, HIV plasma viral load, B12, Venereal Disease Research Laboratory (VDRL), toxic screens for drugs and alcohol, reflex thyroid-stimulating hormone (TSH), urinalysis. Number of participants with a laboratory abnormality meeting specified criteria while on study treatment or during lag time was reported.
Time Frame: Screening up to Week 17
Population: Safety population included all participants who signed the informed consent, had exposure to study drug and had at least one safety assessment. N (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Number; unit: participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 180 | 183
participants | 165 | 170

24. Other Pre Specified Outcome: Number of Participants With Positive Serum and Urine Pregnancy
Description: Serum pregnancy test (regardless of childbearing potential) and urine pregnancy test for all female participants were performed.
Time Frame: Screening for serum pregnancy test, Week 1 for urine pregnancy test
Population: Data for this pre-specified outcome measure was collected and reported in individual participant listings but not statistically summarized for analysis.
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 0 | 0

25. Other Pre Specified Outcome: Number of Participants With Abnormal Physical Examination Findings
Description: A physical examination included an examination of the general appearance, skin, chest, pulses, pulmonary, cardiovascular, head, eyes, ears, nose, throat, abdominal, and extremities.
Time Frame: Screening, Week 8, 17
Population: Safety population included all participants who signed the informed consent, had exposure to open label study drug and had at least one safety assessment. n = participants evaluable for this measure at specified time points for each arm group.
Measure: Number; unit: participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 183 | 192
participants
  Screening: General (n=183, 192) | 16 | 13
  Week 8: General (n=146, 154) | 12 | 7
  Week 17: General (n=170, 174) | 11 | 6
  Screening: Skin (n=183, 192) | 30 | 37
  Week 8: Skin (n=146, 154) | 20 | 20
  Week 17: Skin (n=170, 174) | 21 | 32
  Screening: Chest (n=183, 192) | 6 | 4
  Week 8: Chest (n=146, 154) | 2 | 3
  Week 17: Chest (n=170, 174) | 4 | 2
  Screening: Pulses (n=183, 191) | 3 | 1
  Week 8: Pulses (n=146, 153) | 2 | 1
  Week 17: Pulses (n=170, 174) | 1 | 2
  Screening: Lungs (n=183, 192) | 2 | 6
  Week 8: Lungs (n=146, 154) | 2 | 3
  Week 17: Lungs (n=170, 174) | 3 | 5
  Screening: Heart (n=183, 192) | 3 | 4
  Week 8: Heart (n=146, 154) | 4 | 3
  Week 17: Heart (n=170, 174) | 4 | 3
  Screening: Abdomen (n=183, 192) | 11 | 6
  Week 8: Abdomen (n=146, 154) | 9 | 2
  Week 17: Abdomen (n=170, 174) | 8 | 6
  Screening: Extremities (n=183, 192) | 50 | 46
  Week 8: Extremities (n=146, 154) | 28 | 26
  Week 17: Extremities (n=170, 174) | 29 | 23
  Screening: Head (n=183, 192) | 2 | 5
  Week 8: Head (n=146, 154) | 0 | 2
  Week 17: Head (n=170, 174) | 2 | 2
  Screening: Ears (n=181, 191) | 1 | 3
  Week 8: Ears (n=145, 154) | 0 | 0
  Week 17: Ears (n=170, 174) | 1 | 3
  Screening: Eyes (n=183, 192) | 12 | 7
  Week 8: Eyes (n=146, 154) | 8 | 5
  Week 17: Eyes (n=170, 174) | 9 | 6
  Screening: Nose (n=183, 192) | 0 | 3
  Week 8: Nose (n=146, 154) | 3 | 4
  Week 17: Nose (n=170, 174) | 3 | 1
  Screening: Throat (n=183, 192) | 3 | 3
  Week 8: Throat (n=146, 154) | 4 | 6
  Week 17: Throat (n=170, 174) | 5 | 2

26. Other Pre Specified Outcome: Body Weight
Time Frame: Screening, Week 1, 4, 8, 12, 16, 17
Population: Safety population included all participants who signed the informed consent, had exposure to study drug and had at least one safety assessment. n = participants evaluable for this measure at specified time points for each arm group, respectively.
Measure: Mean (Standard Deviation); unit: kilogram
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 183 | 192
kilogram
  Screening (n=183, 192) | 70.8 (17.7) | 72.0 (17.3)
  Week 1 (n=183, 192) | 71.2 (17.76) | 72.5 (17.84)
  Week 4 (n=158, 169) | 72.6 (19.02) | 71.8 (16.88)
  Week 8 (n=146, 154) | 73.1 (19.35) | 72.1 (17.17)
  Week 12 (n=127, 137) | 74.0 (19.01) | 72.7 (17.20)
  Week 16 (n=170, 176) | 73.6 (18.06) | 72.5 (17.00)
  Week 17 (n=167, 171) | 73.6 (18.13) | 72.6 (16.95)

27. Other Pre Specified Outcome: Sitting Systolic and Diastolic Blood Pressure
Description: Systolic Blood Pressure (SBP) is the blood pressure (pressure exerted by circulating blood on the walls of blood vessels) when heart is contracting; it is the maximum arterial pressure during contraction of left ventricle of heart. Diastolic Blood Pressure (DBP) is the blood pressure (pressure exerted by circulating blood on the walls of blood vessels) when heart is relaxing; it is the minimum arterial pressure during relaxation and dilation of ventricles of heart.
Time Frame: Screening, Week 1, 4, 8, 12, 16, 17
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 183 | 192
millimeter of mercury (mmHg)
  Screening: SBP (n=183, 192) | 121.2 (16.18) | 122.1 (15.02)
  Week 1: SBP (n=183, 192) | 119.9 (14.58) | 120.4 (14.79)
  Week 4: SBP (n=159, 169) | 117.9 (16.42) | 119.8 (15.07)
  Week 8: SBP (n=147, 154) | 118.6 (14.24) | 120.7 (15.18)
  Week 12: SBP (n=127, 137) | 120.2 (15.33) | 121.7 (14.30)
  Week 16: SBP (n=171, 176) | 119.3 (15.71) | 122.9 (13.67)
  Week 17: SBP (n=167, 171) | 120.1 (15.89) | 121.6 (14.35)
  Screening: DBP (n=183, 192) | 78.7 (11.08) | 78.4 (10.84)
  Week 1: DBP (n=183, 192) | 76.9 (10.48) | 77.5 (10.40)
  Week 4: DBP (n=159, 169) | 76.0 (12.01) | 76.5 (10.43)
  Week 8: DBP (n=147, 154) | 76.0 (11.25) | 77.6 (11.27)
  Week 12: DBP (n=127, 137) | 77.5 (10.62) | 78.0 (10.07)
  Week 16: DBP (n=171, 176) | 76.4 (11.07) | 78.1 (9.52)
  Week 17: DBP (n=167, 171) | 76.4 (11.28) | 78.5 (11.48)

28. Other Pre Specified Outcome: Sitting Heart Rate
Time Frame: Screening, Week 1, 4, 8, 12, 16, 17
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 183 | 192
beats per minute (bpm)
  Screening (n=183, 192) | 75.2 (12.44) | 74.6 (11.10)
  Week 1 (n=183, 192) | 76.0 (11.46) | 74.9 (9.27)
  Week 4 (n=159, 169) | 77.5 (10.75) | 77.2 (10.63)
  Week 8 (n=147, 154) | 77.4 (10.52) | 77.1 (10.32)
  Week 12 (n=127, 137) | 78.0 (11.09) | 77.5 (11.09)
  Week 16 (n=171, 176) | 76.2 (11.03) | 76.5 (11.17)
  Week 17 (n=167, 171) | 76.0 (10.91) | 76.2 (10.35)

29. Other Pre Specified Outcome: Number of Participants With Neurological Examination Findings
Description: A neurological examination consisted of examination of the mental state, cranial nerve function, motor function (reflexes of patellar, achilles, biceps, babinski and coordination) and sensory function (sharp sensation of dorsal surface of right and left great toe, light touch of lower extremities [LE], right and left first metatarsal joint position sense, and vibration sensation [vibration is felt for < 6 seconds = markedly diminished, 6 to 10 seconds = mild loss, > 10 seconds = normal]).
Time Frame: Screening
Population: as for outcome 22
Measure: Number; unit: participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 183 | 192
participants
  Cranial Nerve Function: Missing | 1 | 0
  Cranial Nerve Function: Normal | 178 | 192
  Cranial Nerve Function: Abnormal | 4 | 0
  Cranial Nerve Function: Not Done | 0 | 0
  Coordination, Gait: Missing | 1 | 1
  Coordination, Gait: Normal | 169 | 181
  Coordination, Gait: Not Evaluable | 2 | 2
  Coordination, Gait: Mild Ataxia | 7 | 7
  Coordination, Gait: Moderate Ataxia | 3 | 1
  Coordination, Gait: Severe Ataxia | 1 | 0
  Coordination, Romberg Test: Missing | 1 | 0
  Coordination, Romberg Test: Normal | 174 | 188
  Coordination, Romberg Test: Abnormal | 6 | 2
  Coordination, Romberg Test: Not Done | 2 | 2
  Reflexes, Left Patellar: Missing | 1 | 0
  Reflexes, Left Patellar: None/Absent | 7 | 13
  Reflexes, Left Patellar: Normal | 124 | 130
  Reflexes, Left Patellar: Not Done | 0 | 0
  Reflexes, Left Patellar: Hypoactive (Diminished) | 43 | 41
  Reflexes, Left Patellar: Hyperactive (More Brisk) | 8 | 8
  Reflexes, Left Patellar: Clonus (Very Intense) | 0 | 0
  Reflexes, Right Patellar: Missing | 1 | 0
  Reflexes, Right Patellar: None/Absent | 8 | 13
  Reflexes, Right Patellar: Normal | 124 | 129
  Reflexes, Right Patellar: Not Done | 1 | 0
  Reflexes, Right Patellar: Hypoactive (Diminished) | 42 | 41
  Reflexes, Right Patellar: Hyperactive (More Brisk) | 7 | 9
  Reflexes, Right Patellar: Clonus (Very Intense) | 0 | 0
  Reflexes, Left Achilles: Missing | 1 | 0
  Reflexes, Left Achilles: None/Absent | 92 | 100
  Reflexes, Left Achilles: Normal | 14 | 13
  Reflexes, Left Achilles: Not Done | 0 | 0
  Reflexes, Left Achilles: Hypoactive (Diminished) | 73 | 78
  Reflexes, Left Achilles: Hyperactive (More Brisk) | 3 | 1
  Reflexes, Left Achilles: Clonus (Very Intense) | 0 | 0
  Reflexes, Right Achilles: Missing | 1 | 0
  Reflexes, Right Achilles: None/Absent | 90 | 100
  Reflexes, Right Achilles: Normal | 14 | 9
  Reflexes, Right Achilles: Not Done | 0 | 0
  Reflexes, Right Achilles: Hypoactive (Diminished) | 75 | 82
  Reflexes, Right Achilles: Hyperactive (More Brisk) | 3 | 1
  Reflexes, Right Achilles: Clonus (Very Intense) | 0 | 0
  Reflexes, Right Biceps: Missing | 1 | 0
  Reflexes, Right Biceps: None/Absent | 1 | 2
  Reflexes, Right Biceps: Normal | 166 | 178
  Reflexes, Right Biceps: Not Done | 3 | 2
  Reflexes, Right Biceps: Hypoactive (Diminished) | 8 | 7
  Reflexes, Right Biceps: Hyperactive (More Brisk) | 4 | 3
  Reflexes, Right Biceps: Clonus (Very Intense) | 0 | 0
  Reflexes, Left Biceps: Missing | 1 | 0
  Reflexes, Left Biceps: None/Absent | 1 | 2
  Reflexes, Left Biceps: Normal | 169 | 180
  Reflexes, Left Biceps: Not Done | 2 | 1
  Reflexes, Left Biceps: Hypoactive (Diminished) | 7 | 6
  Reflexes, Left Biceps: Hyperactive (More Brisk) | 3 | 3
  Reflexes, Left Biceps: Clonus (Very Intense) | 0 | 0
  Mental State: Missing | 3 | 0
  Mental State: Normal | 179 | 192
  Mental State: Abnormal | 1 | 0
  Mental State: Not Done | 0 | 0
  Sensory Function, Right Great Toe: Missing | 1 | 0
  Sensory Function, Right Great Toe: Absent | 63 | 57
  Sensory Function, Right Great Toe: Diminished | 99 | 114
  Sensory Function, Right Great Toe: Normal | 5 | 7
  Sensory Function, Right Great Toe: Increased | 15 | 14
  Sensory Function, Left Great Toe: Missing | 1 | 0
  Sensory Function, Left Great Toe: Absent | 61 | 58
  Sensory Function, Left Great Toe: Diminished | 102 | 112
  Sensory Function, Left Great Toe: Normal | 5 | 8
  Sensory Function, Left Great Toe: Increased | 14 | 14
  Sensory Function-Light Touch, LE: Missing | 2 | 3
  Sensory Function-Light Touch, LE: Not Done | 7 | 6
  Sensory Function-Light Touch, LE: Unable to Detect | 39 | 48
  Sensory Function-Light Touch, LE: Hyposensitivity | 99 | 102
  Sensory Function-Light Touch, LE: Normal Sensation | 28 | 25
  Sensory Function-Light Touch, LE: Hypersensitivity | 8 | 8
  Sensory Function, Right Metatarsal Sense: Missing | 1 | 0
  Sensory Function, Right Metatarsal Sense: Normal | 129 | 143
  Sensory Function, Right Metatarsal Sense: Abnormal | 52 | 47
  Sensory Function, Right Metatarsal Sense: Not Done | 1 | 2
  Sensory Function, Left Metatarsal Sense: Missing | 1 | 0
  Sensory Function, Left Metatarsal Sense: Normal | 129 | 143
  Sensory Function, Left Metatarsal Sense: Abnormal | 51 | 46
  Sensory Function, Left Metatarsal Sense: Not Done | 2 | 3
  Vibration Sensation: Missing | 2 | 2
  Vibration Sensation: Not Done | 1 | 1
  Vibration Sensation: Absent | 27 | 24
  Vibration Sensation: Markedly Diminished | 42 | 52
  Vibration Sensation: Mild Loss | 86 | 79
  Vibration Sensation: Normal | 25 | 34
  Reflexes, Right Babinski: Missing | 1 | 0
  Reflexes, Right Babinski: Not Evaluable | 3 | 6
  Reflexes, Right Babinski: Absent | 173 | 180
  Reflexes, Right Babinski: Present | 6 | 6
  Reflexes, Left Babinski: Missing | 1 | 0
  Reflexes, Left Babinski: Not Evaluable | 3 | 6
  Reflexes, Left Babinski: Absent | 173 | 180
  Reflexes, Left Babinski: Present | 6 | 6

30. Other Pre Specified Outcome: Number of Participants Who Met Mini-International Neuropsychiatric Interview (MINI) Criteria
Description: MINI: short structured clinical interview to make diagnoses of psychiatric disorders according to Diagnostic and Statistical Manual of Mental Disorders-IV (DSM-IV) or International Classifications of Disease-10 (ICD-10). In the MINI Modules, participants were asked a series of Yes/No questions.
Time Frame: Screening
Population: as for outcome 24
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 0 | 0

31. Other Pre Specified Outcome: Number of Participants With Response to Sheehan-Suicidality Tracking Scale (S-STS) Mapped to the Columbia Classification Algorithm of Suicide Assessment (C-CASA) Categories
Description: S-STS:8-item clinician/participant administered prospective rating scale to assess TE suicidal(Su) ideation(ID),behavior(BHV).Items 1a,2-6,7a,8 scored on 5-point Likert scale 0(not at all) to 4(extremely). Items 1,1b,7 require yes/no response. S-STS total score range 0-30. Lower score=reduced Su tendency. Responses on S-STS were mapped to Columbia Classification Algorithm of Suicide Assessment(C-CASA) as 1:Completed Su; 2: Su attempt; 3: Preparatory acts; 4: Su ID; 5: Self-injurious (SI) BHV, intent unknown; 6: Not enough information; 7: SI BHV, no Su intent; 8: Other, no deliberate self harm.
Time Frame: Screening, Post-Baseline (Week 4 up to Week 17)
Population: as for outcome 26
Measure: Number; unit: participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 183 | 192
participants
  Screening: Su Attempt (n=183, 192) | 5 | 8
  Screening: Preparatory Acts (n=183, 192) | 5 | 8
  Screening: Su ID (n=183, 192) | 28 | 37
  Screening: SI BHV, no Su intent (n=183, 192) | 4 | 4
  Post-Baseline: Completed Suicide (n=178, 185) | 0 | 0
  Post-Baseline: Su Attempt (n=178, 185) | 0 | 1
  Post-Baseline: Preparatory Acts (n=178, 185) | 0 | 2
  Post-Baseline: Su ID (n=178, 185) | 5 | 11
  Post-Baseline: SI BHV, no Su intent (n=178, 185) | 0 | 0

32. Other Pre Specified Outcome: Number of Participants With Response to Patient Health Questionnaire-8 (PHQ-8)
Description: PHQ-8: 8-item self-administered validated subset of PHQ-9, which comprises first 8 items of measure. Participant rated "Over past 2 weeks, how often bothered by any of following problems?": little interest in doing things(1); feeling down(2); trouble falling or staying asleep/sleeping too much(3); feeling tired(4); poor appetite/overeating(5); feeling bad about self(6); trouble concentrating(7); moving or speaking slowly or being so fidgety/moving around more than usual (8). Each item scored on scale of 0(not at all)-3(nearly every day). Total score range: 0-24, higher score=greater severity.
Time Frame: Screening
Population: as for outcome 19
Measure: Number; unit: participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 183 | 192
participants
  Little Interest: Not at All (n=183, 192) | 77 | 89
  Little Interest: Several Days (n=183, 192) | 63 | 72
  Little Interest: > 1/2 Days (n=183,192) | 23 | 20
  Little Interest: Nearly Every Day (n=183, 192) | 20 | 11
  Feeling Down: Not at All (n=183, 192) | 105 | 109
  Feeling Down: Several Days (n=183, 192) | 61 | 59
  Feeling Down: > 1/2 Days the Days (n=183, 192) | 13 | 12
  Feeling Down: Nearly Every Day (n=183, 192) | 4 | 12
  Trouble With Sleep: Not at All (n=182, 192) | 63 | 68
  Trouble With Sleep: Several Days (n=182, 192) | 69 | 86
  Trouble With Sleep: > 1/2 Days (n=182, 192) | 26 | 22
  Trouble With Sleep: Nearly Every Day (n=182, 192) | 24 | 16
  Feeling Tired: Not at All (n=183, 192) | 57 | 56
  Feeling Tired: Several Days (n=183, 192) | 87 | 100
  Feeling Tired: > 1/2 Days (n=183, 192) | 27 | 29
  Feeling Tired: Nearly Every Day (n=183, 192) | 12 | 7
  Poor Appetite/Overeat: Not at All (n=183, 192) | 99 | 116
  Poor Appetite/Overeat: Several Days (n=183, 192) | 53 | 56
  Poor Appetite/Overeat: > 1/2 Days (n=183, 192) | 21 | 15
  Poor Appetite/Overeat: Nearly Everyday (n=183,192) | 10 | 5
  Feeling Bad About Self: Not at All (n=183, 192) | 124 | 138
  Feeling Bad About Self: Several Days (n=183, 192) | 41 | 43
  Feeling Bad About Self: > 1/2 Days (n=183, 192) | 12 | 6
  Feeling Bad About Self: Nearly Everyday(n=183,192) | 6 | 5
  Trouble Concentrating: Not at All (n=183, 192) | 131 | 140
  Trouble Concentrating: Several Days (n=183, 192) | 35 | 33
  Trouble Concentrating: > 1/2 Days (n=183, 192) | 11 | 13
  Trouble Concentrating: Nearly Everyday (n=183,192) | 6 | 6
  Move-Speak Slow/Fidgety: Not at All (n=183,192) | 144 | 143
  Move-Speak Slow/Fidgety:Several Days(n=183,192) | 23 | 33
  Move-Speak Slow/Fidgety: >1/2 Days (n=183, 192) | 10 | 10
  Move-Speak Slow/Fidgety:Nearly Everyday(n=183,192) | 6 | 6

33. Secondary Outcome: Diagnostic Neuropathy Assessment
Time Frame: Screening
Population: Data were not collected since this was a screening tool for investigators and there was no analysis planned for this measure.
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Pregabalin | Placebo
Serious Adverse Events (participants affected / at risk) | 7/183 | 7/192
Other Adverse Events (participants affected / at risk) | 64/183 | 47/192
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=183) | Placebo (N=192)
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Gallbladder disorder (Hepatobiliary disorders) | 0 | 1
Perineal abscess (Infections and infestations) | 1 | 0
Pneumocystis jiroveci pneumonia (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Demyelinating polyneuropathy (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=183) | Placebo (N=192)
Influenza (Infections and infestations) | 17 | 12
Dizziness (Nervous system disorders) | 25 | 10
Headache (Nervous system disorders) | 25 | 26
Somnolence (Nervous system disorders) | 13 | 4

LIMITATIONS AND CAVEATS:
Based on Data Monitoring Committee (DMC) interim efficacy analysis results indicating a low probability for success, the study was terminated on April 2, 2012; the termination was unrelated to any safety findings that could impact participant health.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.